CLINICAL TRIAL: NCT01191476
Title: A Prospective, Randomized, Open-label Multicenter Study Comparing the Pharmaceutical Economics and Effectiveness of Sevoflurane With Low Fresh Gas Flow Balanced Anesthesia, Propofol Target Controlled Infusion Anesthesia and Propofol Induction Sevoflurane Maintenance Anesthesia in Laparoscopic Surgeries in China
Brief Title: Compare Pharmaceutical Economics and Efficacy of Sevoflurane With Low Fresh Gas Flow Balanced Anesthesia, Propofol Target Controlled Infusion Anesthesia and Propofol Induction Sevoflurane Maintenance Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Rundo International Pharmaceutical Research & Development Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R12-564
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-05

CONDITIONS: Elective Laparoscopic Surgery
Keywords: Sevoflurane; Propofol; Economics; Pharmaceutical; Chinese
MeSH Terms: interventions — Maintenance; Sevoflurane; Neoadjuvant Therapy; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane (Active Comparator): Subjects received sevoflurane, a inhalational (volatile) anesthetic, which was administered for induction and maintenance of general anesthesia. Inhalational induction was induced via vital capacity induction at 8% and maintained at 0.8-1.5 minimum alveolar concentration (MAC).
  Interventions: Drug: Sevoflurane Inhalational Induction and Maintenance
- Propofol (Active Comparator): Subjects received propofol, an intravenous (IV) anesthetic, which was administered for induction and maintenance of general anesthesia.
  Interventions: Drug: Propofol Target Controlled Infusion for Induction and Maintenance
- Propofol Induction and Sevoflurane Maintenance (Active Comparator): Subjects received a bolus dose of propofol of 1.5 mg/kg administered for IV induction followed by sevoflurane at 0.8-1.5 MAC for maintenance anesthesia.
  Interventions: Drug: Propofol Target Controlled Infusion for Induction and Sevoflurane Inhalation for Maintenance

INTERVENTIONS:
Drug: Sevoflurane Inhalational Induction and Maintenance — Sevoflurane was administered at a concentration of 8% via vital capacity induction and sevoflurane 0.8-1.5 minimum alveolar concentration (MAC) with a rate of 1 L/min fresh gas flow for maintenance.
  Other Names: ABT-941; sevoflurane; Ultane; Sevorane; Sevofrane
  Arms: Sevoflurane
Drug: Propofol Target Controlled Infusion for Induction and Maintenance — Propofol IV 4 ug/mL was administered with target controlled infusion (TCI) for induction and propofol 3 to 6 ug/mL was administered with TCI for maintenance.
  Other Names: Propofol
  Arms: Propofol
Drug: Propofol Target Controlled Infusion for Induction and Sevoflurane Inhalation for Maintenance — Propofol was administered as a bolus IV dose of 1.5 mg/kg for induction at a rate of 40 mg/10 seconds. During maintenance, a sevoflurane concentration of 0.8-1.5 minimal alveolar concentration (MAC) was administered at a rate of 1 L/min fresh gas flow.
  Other Names: ABT-941; sevoflurane; Ultane; Sevorane; Sevofrane
  Arms: Propofol Induction and Sevoflurane Maintenance

SUMMARY:
This study is being performed to compare the cost of anesthetic techniques with sevoflurane (low fresh gas flow balanced anesthesia) versus propofol (target controlled infusion [TCI]) versus propofol induction and sevoflurane maintenance anesthesia in subjects undergoing elective laparoscopic surgery with predicted anesthesic use between 1 and 3 hour duration.

DETAILED DESCRIPTION:
Three hundred thirty-six subjects were enrolled in this study. Two subjects, one treated with propofol for induction and maintenance and one treated with propofol for induction and sevoflurane for maintenance are not included in the study participation since no information was available for these two subjects.

ELIGIBILITY:
Inclusion Criteria

1. Men or women, aged from 18 to 65
2. ASA (American Society of Anesthesiologists) physical status (a requirement of the subject's physical status): I or II
3. Body mass index (weight/height^2) from 16 to 30 kg/m^2
4. Elective laparoscopic surgery requiring general anesthesia managed with endotracheal intubation
5. Duration of anesthesia use will be greater than or equal to 1 hour, but less than 3 hours in length.

Exclusion Criteria

1. Hypersensitivity or unusual response to any halogenated anesthetics.
2. History of significant cardiovascular, pulmonary, hepatic, renal, central nervous system or muscular disease.
3. Pre-operative cognitive dysfunction or disabling neuropsychiatric disorders.
4. Need for emergency surgery or surgery requiring additional regional anesthetic techniques.
5. Need for intracranial surgery, cardio-surgery or thoracic surgery.
6. Subjects inability to cooperate with the anesthetist before administration of the anesthetic agent.
7. Personal or familial history of malignant hyperthermia.
8. Females who are either pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Kang, MD, Study Director — Abbott
Locations (4):
- China (4):
  - Site Reference ID/Investigator# 41983, Beijing
  - Site Reference ID/Investigator# 41932, Chengdu
  - Site Reference ID/Investigator# 41985, Guangzhou
  - Site Reference ID/Investigator# 41984, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects between the ages of 18 and 65 were recruited from 4 hospitals in 4 cities in China. They were required to have elective laparoscopic, in-patient surgery with a predicted anesthetic duration between 1 to 3 hours. Subjects with ASA physical status I or II were enrolled and were to have had the ability to provide informed consent.
Pre-assignment Details: The study was a prospective, randomized (1:1:1), open-label, multi-center study comparing the cost of inhalational anesthesia with sevoflurane to intravenous (IV) anesthesia with propofol, or propofol for induction and sevoflurane for maintenance of anesthesia. The full analysis set was used for determination of all primary and secondary endpoints.
Groups:
- Sevoflurane: Inhalational induction and maintenance anesthesia with sevoflurane.
- Propofol: Target controlled infusion anesthesia with propofol for induction and maintenance.
- Propofol Induction Sevoflurane Maintenance: Propofol induction and sevoflurane maintenance anesthesia.
Period: Overall Study
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Started | 112 | 111 (Data was not collected for 1 subject for baseline characteristics or the full analysis set.) | 111 (Data was not collected for 1 subject for baseline characteristics or the full analysis set.)
Completed | 109 | 107 | 111
Not Completed | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance | Total
Number analyzed (Participants) | 112 | 111 | 111 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 112 | 111 | 111 | 334
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.29 (12.15) | 43.26 (12.05) | 42.51 (11.81) | 42.71 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 87 | 271
  Male | 20 | 19 | 24 | 63
Region of Enrollment [Number; unit: participants]
  China | 112 | 111 | 111 | 334

OUTCOME MEASURES:

1. Primary Outcome: Cost of Volatile Induction and Maintenance Anesthesia (VIMA) With Sevoflurane, Total Intravenous Anesthesia (TIVA) With Propofol, or Intravenous Induction With Propofol and Inhalational Maintenance With Sevoflurane
Description: [Cost of VIMA = unit price of sevoflurane X used volume of sevoflurane];
  [Cost of TIVA = unit price of propofol X total volume of propofol in the syringe];
  [Cost of Propofol Induction and Sevoflurane Maintenance = unit price of propofol X total volume of propofol in the syringe + unit price of sevoflurane X volume of sevoflurane in the syringe].
  The total volume of propofol in the syringe was calculated, even if all the anesthetic was not used, because it could not be reused.
Time Frame: Anesthetic Duration between 1 to 3 Hours
Population: The full analysis set was used for the determination of cost of anesthesia.
Measure: Mean (Standard Deviation); unit: Yuan
Groups:
- Sevoflurane: Inhalational sevoflurane for induction and maintenance of anesthesia
- Propofol: IV Propofol for induction and maintenance of anesthesia
- Propofol Induction Sevoflurane Maintenance: Propofol bolus for IV induction and sevoflurane for maintenance of anesthesia
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Number analyzed (Participants) | 112 | 111 | 111
Yuan | 380.78 (108.53) | 548.52 (195.14) | 269.40 (74.04)

2. Secondary Outcome: Time to Loss of Consciousness
Description: Loss of consciousness was measured from the time the anesthetic was administered until loss of consciousness (no response to command) occurred. Inhalational induction was induced with sevoflurane via vital capacity induction at 8%. Intravenous induction was induced with propofol at 4 µg/mL via target controlled infusion (TCI). In subjects who received both anesthetic agents, a bolus dose of propofol 1.5 mg/kg was used for induction.
Time Frame: Up to 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Number analyzed (Participants) | 112 | 111 | 111
seconds | 48.54 (22.77) | 100.32 (55.15) | 68.76 (34.96)

3. Secondary Outcome: Time to Eye Opening
Description: Measured from the time sevoflurane or propofol administration was stopped until the subject's eyes were opened. The investigator tapped the subject on the forehead or shoulder after anesthesia was stopped and asked them to open their eyes. This process was repeated approximately every minute until eye opening occurred.
Time Frame: Every minute after anesthesia was stopped until the subjects' eyes opened
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Number analyzed (Participants) | 112 | 111 | 111
Minutes | 8.38 (3.66) | 9.79 (6.92) | 8.69 (3.50)

4. Secondary Outcome: Time to Extubation
Description: Time to extubation was measured from the time sevoflurane or propofol administration was stopped until tracheal extubation occurred. Criteria to determine extubation included a train of four stimulus > 0.9 (a method to measure the magnitude and type of neuromuscular block, a ratio of the fourth response to the first one), a tidal volume > 5 mL/kg, minute ventilation > 3 L, a respiratory rate of > 10 breaths/minute, an end tidal carbon dioxide < 45 mmHg, and eye opening has occurred.
Time Frame: Every minute after anesthesia was stopped until extubation occurred
Population: Measurement
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Propofol Induction and Sevoflurane Maintenance: Propofol bolus for IV induction and sevoflurane for maintenance of anesthesia
Arm/Group | Sevoflurane | Propofol | Propofol Induction and Sevoflurane Maintenance
Number analyzed (Participants) | 112 | 111 | 111
Minutes | 9.69 (3.84) | 11.32 (6.91) | 9.79 (3.52)

5. Secondary Outcome: Time to Orientation
Description: Time to orientation was measured from the time sevoflurane or propofol administration was stopped until orientation (able to state their name and date of birth).
Time Frame: Every minute after anesthesia was stopped until orientation occurred
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Number analyzed (Participants) | 112 | 111 | 111
Minutes | 13.97 (6.73) | 17.64 (12.45) | 14.95 (6.39)

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time study drug was administered until 30 days after the study drug treatment was completed. Serious adverse events were collected from the time the subject signed the informed consent form.
Arm/Group | Sevoflurane | Propofol | Propofol Induction Sevoflurane Maintenance
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/111 | 0/111
Other Adverse Events (participants affected / at risk) | 5/112 | 4/111 | 5/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sevoflurane (N=112) | Propofol (N=111) | Propofol Induction Sevoflurane Maintenance (N=111)
bradycardia (Cardiac disorders) | 3 | 0 | 1
diastolic blood pressure decreased (Investigations) | 0 | 0 | 1
hypotension (Vascular disorders) | 3 | 2 | 2
Movement Disorder (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.